CLINICAL TRIAL: NCT02020200
Title: A Crossover Study on the Effect of Methylphenidate (MPH) on Cognitive Abilities of Adults With Bipolar Disorder (BD), During Remission or Depressed State, Compared With Healthy Adults and Adults With Attention Deficit Hyperactivity Disorder (ADHD).
Brief Title: The Effect of Methylphenidate on Cognitive Abilities of Adults With Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 0021-12-SHA
Record Dates: First submitted 2013-12-14; First posted 2013-12-24 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: BD
Keywords: Bipolar Disorder; Methylphenidate; Cognitive Function
MeSH Terms: conditions — Bipolar Disorder | interventions — 5,10-dihydro-5-methylphenazine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- MPH or Placebo (Experimental): MPH dosage will be determined according to participants' body weight: dosage: 10 mg in case weight<40 kg; 30 mg in case weight>90 kg; otherwise 20 mg. Both participants and investigators will be blinded to when participant receives MPH or Placebo.
  Interventions: Drug: MPH; Drug: Placebo

INTERVENTIONS:
Drug: MPH — MPH dosage will be determined according to participants' body weight: dosage: 10 mg in case weight<40 kg; 30 mg in case weight>90 kg; otherwise 20 mg.
  Other Names: Ritalin
Drug: Placebo

SUMMARY:
The purpose of the study is to explore the effect of MPH on working memory, attention and decision making in adults with BD in remission or in depressed state. The results will be compared to findings in healthy adults and adults with ADHD. The investigators hypothesize that MPH will incur improved performance in all measures.

DETAILED DESCRIPTION:
Following a detailed explanation about the trial and after obtaining informed consent from candidates, subjects will be asked to arrive at the cognitive laboratory at Shalvata MHC twice. Visits will include performance of computerized cognitive and decision making tasks, as well as two creativity tasks after the consumption of MPH or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew Speakers
* Age 21-50
* Diagnosis of BD I or II (296.7 and 296.89 classifications in the DSM-IV-TR), according to medical records. Diagnosis will be confirmed by a psychiatrist during screening process using the Structured Clinical Interview for DSM-IV-TR (SCID).

Exclusion Criteria:

* Diagnosis of a clinical disorder other than BD or ADD/ADHD which may impair performance on tasks used in the study.
* BD patients diagnosed with an acute manic episode at screening, as established by YMRS>8. It will also be required that 3 months have elapsed since the latest manic state, according to the patients' history.
* Participants for whom there exists a contra-indication for consuming Ritalin.
* Pregnancy or current breastfeeding; Female participants will be asked to report whether they are pregnant or currently nursing and if so, they will be excluded from the study.
* Drug use in the previous 6 weeks according to participants' self report
* Electroconvulsive therapy (ECT) in the previous 6 months

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive function. | Within 4 hours of intervention.
  Cognitive function will be measured by scores on several computerized neuro-psychological and decision making tasks: digit-span task, spatial working memory task, raven's progressive matrices, test of variable attention and the Iowa gambling task.

SECONDARY OUTCOMES:
Creativity abilities. | Within 4 hours of intervention.
  Creativity will be measured by scores on two tests: the alternative use task and two subsets of the Torrance tests for creative thinking.

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, PhD, Principal Investigator — Shalavata MHC
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel